CLINICAL TRIAL: NCT06971783
Title: Effect of an Experimental Gel Based on Acmella Oleracea Extract Associated or Not With Fluoride on Dentin Hypersensitivity: a Randomized Clinical Study
Brief Title: Effect of an Experimental Gel Based on Acmella Oleracea Extract Associated or Not With Fluoride on Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Professor of the Graduate Program in Dentistry at the Federal University of Pará, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7.513.177
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dentin Desensitizers; Non-carious Cervical Lesions; Dentin Hypersensitivity
Keywords: Acmella oleracea; Spilanthol; Dentin hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Fluorides

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT group: negative control group (Placebo Comparator): the group will receive the application of gel without active ingredient
  Interventions: Other: CT- control group
- NP Group - Potassium nitrate associated with 2% Fluoride (Active Comparator): the group will receive the application of gel containing potassium nitrate
  Interventions: Other: NP- Potassium nitrate gel
- Group AO - Acmella Oleracea extract gel (Experimental): the group will receive the application of gel containing Acmella Oleracea Extract Gel
  Interventions: Other: AO - Acmella Oleracea Extract Gel
- AF Group - Acmella Oleracea extract gel associated with Fluoride. (Experimental): the group will receive the application of gel containing Acmella Oleracea Extract Gel associated with fluoride
  Interventions: Other: AF - Gel of Acmella Oleracea extract associated with Fluoride.

INTERVENTIONS:
Other: CT- control group — will receive the application of a placebo gel (without active ingredient), under the same conditions described for the experimental gel.
  Arms: CT group: negative control group
Other: NP- Potassium nitrate gel — The gels will be applied to the sensitive lesions according to the experimental group and will be rubbed for 20 seconds using a microbrush, remaining on the lesions for 10 minutes.
  Arms: NP Group - Potassium nitrate associated with 2% Fluoride
Other: AO - Acmella Oleracea Extract Gel — The Acmella oleracea gel will be applied to sensitive lesions and rubbed for 20 seconds with the aid of a microbrush, remaining on the lesions for 10 minutes.
  Arms: Group AO - Acmella Oleracea extract gel
Other: AF - Gel of Acmella Oleracea extract associated with Fluoride. — The Acmella oleracea gel associated with fluoride will be applied to sensitive lesions and rubbed for 20 seconds with the aid of a microbrush, remaining on the lesions for 10 minutes.
  Arms: AF Group - Acmella Oleracea extract gel associated with Fluoride.

SUMMARY:
This randomized, single-blind, placebo-controlled clinical trial aims to evaluate the effect of an experimental gel based on Acmella oleracea (jambú) extract, associated or not with fluoride, in reducing dentin hypersensitivity (DH) in non-carious cervical lesions. The volunteers were randomized into 4 groups according to the treatments applied: CT (control), NP (potassium nitrate), AO (Acmella oleracea) and AF (Acmella oleracea associated with fluoride). Prophylaxis with pumice stone and water was performed on the previously selected teeth and, subsequently, the gels were applied to the cervical region with a microbrush, rubbed for 10 seconds, and remained on the tooth surface for 10 minutes. Three gel application sessions were performed, with 1-week interval between them. The DH evaluation was performed at four time points: baseline (before the first session), T1 (before the second session), T2 (before the third session) and T3, one week after the final application of the products.

DETAILED DESCRIPTION:
Initially, all volunteers will undergo prophylaxis with pumice and water and will receive an oral hygiene kit containing a soft-bristled toothbrush, dental floss, and their assigned toothpaste, along with oral hygiene instructions. Relative isolation with cotton rolls will be performed in the region of the sensitive lesions, followed by the application of the gel corresponding to the participant's group (CT, NP, AO, AF). All gels will be applied in the same manner, using a microbrush applicator. After being rubbed for 20 seconds on each tooth, the gel will remain on the tooth surface for 10 minutes. At the end of this period, the gel will be removed using gauze and thoroughly rinsed. Three clinical sessions will be conducted, with one-week intervals between them.

ELIGIBILITY:
Inclusion Criteria:

* Presence of non-carious cervical lesions with sensitivity and up to 2 mm in depth
* Miller Class I gingival recession
* Lesions located on the buccal surface of the teeth
* Score ≥ 4 on the Visual Analog Scale (VAS) after tactile and evaporative stimuli
* Healthy periodontal condition
* No other conditions that could explain dentin hypersensitivity
* Good general physical health
* No eating disorders or high-acid diets
* Occlusal stability

Exclusion Criteria:

* Presence of restorations in the hypersensitive areas
* Presence of dental caries, pulpitis, or periodontal pockets
* Enamel cracks
* Systemic diseases
* Continuous use of antibiotics, anti-inflammatory drugs, analgesics, or corticosteroids
* Professional desensitizing treatment received within the three months prior to study recruitment
* Pregnancy or breastfeeding Ongoing orthodontic treatment
* Dental prostheses that may interfere with the assessment of hypersensitivity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
sensitivity assessment | 30 days
  Dentin hypersensitivity (DH) will be assessed at four time points: baseline (immediately before the first session), T1 (immediately before the second session), T2 (immediately before the third session), and T3 (one week after the final application of the products). DH will be evaluated using the Visual Analog Scale (VAS). This scale consists of a 10 cm horizontal line with scores of 0 and 10 at each end, where 0 indicates no sensitivity and 10 indicates severe dental sensitivity. Patients will be instructed to draw a vertical line along the horizontal scale to indicate the intensity of their dental sensitivity on the day of assessment.The distance from the zero end to the patient's mark will be measured using a millimeter ruler. These data will be recorded and tabulated for subsequent analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, Principal Investigator — universidade federal do pará
Locations (1):
- Universidade Federal Do Para, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No